CLINICAL TRIAL: NCT04829448
Title: The Influence of a Protein Nutrition Beverage on Exercise-based Rehabilitation Outcomes in Individuals with Spine Pain.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Protein product reconfiguration
Sponsor: Kamshad Raiszadeh, MD (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor-Investigator, Kamshad Raiszadeh, MD, Chairman, Cheif Medical Officer, SpineZone Medical Fitness, Inc
Organization: SpineZone Medical Fitness, Inc (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Protein and Exercise Outcomes
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Low Back Pain
Keywords: Protein Supplement; Exercise-based Rehabilitation
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Protein Intervention Group (Experimental): Patients who receive the protein nutritional supplement as part of their prescribed exercise-based rehabilitation program.
  Interventions: Dietary Supplement: Protein supplement
- Control Group (No Intervention): Patients who receive the prescribed exercise-based rehabilitation program, without protein supplement.

INTERVENTIONS:
Dietary Supplement: Protein supplement — Protein supplement equivalent to Metagenics Ultrameal
  Arms: Protein Intervention Group

SUMMARY:
SpineZone is an innovative physical therapy program with its focus on treatment of cervical, thoracic, and lumbar conditions through the use of a multi-disciplinary, technology enabled platform. Standard physical therapy modalities including exercise-based rehabilitation as well as patient education on a healthy lifestyle (sleep, nutrition, posture) are employed as part of the standard treatment. As nutrition is a key element in modulating muscle growth and function in response to exercise, providing patients with appropriate access to nutritional supplements that meet the metabolic demands of our exercise program are potentially important to our clinical outcomes.

DETAILED DESCRIPTION:
Low back pain manifests itself clinically with pain, loss of strength, difficulty with normal posture, and decreased range of motion. In as many as 60-85% cases, LBP will become a chronic condition, requiring long term care, and even surgery.

Conservative therapy is typically administered until it's no longer a viable option, after which surgical options are considered. Conservative therapy includes physical therapy, medication, steroid injections etc. Physical therapy and exercises are especially central to conservative therapy. Numerous exercise and therapy protocols have been designed with the goal to improve low back muscle strength, thereby alleviating symptoms, and potentially underlying cause of the pathology.

As nutrition is a key element in modulating muscle growth and function in response to exercise, providing patients with appropriate access to nutritional supplements that meet the metabolic demands of our exercise program are potentially important to our clinical outcomes.

The project specifically aims to assess the effect of ensuring adequate nutritional availability of protein, as protein shake, as part of their standard care for treatment of low back pain typically 4-12 weeks duration. In this experiment, we will compare muscle structure and health and correlate improvements with patient-specific characteristics such as demographics, medical history, medication usage, treatment expectations, and symptom severity. Subsequently, this information will enable us to gain valuable insight into physiological response of pathological tissue, and potentially, develop optimal exercise plans to maximally benefit these patients.

AIMS OF THE STUDY

* To evaluate the adherence and compliance of patients taking a protein nutritional supplement in this patient population.
* To evaluate the effectiveness of protein nutritional supplementation on improving clinical outcomes.
* Identify patients (based on patient specific predictors who are most likely to succeed with the addition of nutritional supplementation. The goal of this project is to assess the impact of a nutritional protein supplement on clinical outcomes in individuals with spine pain.

RESEARCH PARTICIPANTS We will recruit up to 100 individuals with LBP of > 3months duration that have been identified by the care providers (ie. Primary care physical, orthopaedic surgeon, or other) to be appropriate and safe for participation in a physical rehabilitation program with nutritional supplementation at SpineZone.

Upon initial evaluation at the SpineZone clinic with a Physical Therapist, participants will be offered the opportunity participate in the study and may receive the protein supplement as part of their standard care. Potentially interested patients will be screened by inclusion and exclusion criteria and as such, written informed consent will be obtained from each patient.

Patients will then be randomly assigned to the treatment (protein supplement) or control group (no protein supplement) and commence their prescribed rehabilitation treatment as per therapist recommendation. Individuals in the randomly assigned supplementation group will be provided the supplement and will be instructed on its use (dosage and frequency).

CONSENT All guidelines for proper consenting will be observed. Consenting will be done in a private room prior to any procedures being performed. Patients will be given ample time to review the document and ask questions. All study procedures will be thoroughly explained and all questions will be answered. Patients will not be placed under any pressure to participate in the study. Consent forms will be obtained by the investigators of the study and/or the study coordinator in the SpineZone clinics.

Withdrawal from the study: If the patient decides at any point to withdraw from the study, they can do so without any of the benefits to which they are entitled changing.

RISK/BENEFITS RATIO The risks to the patients will be minimal. Although there is, future patients may benefit from improvements to surgical procedures and more effective rehabilitation programs which will be derived from patient outcomes.

DATA PRIVACY AND CONFIDENTIALITY A confidentiality breach is a risk associated with data review research; however every measure will be instituted to ensure that patient information is kept confidential. Data analysis worksheets will be kept separate from EMR records. No subject public health information will be collected or shared.

ELIGIBILITY:
Inclusion Criteria:

* Seeking treatment for spinal conditions, pain or for the prevention of future injury
* Ability to consume protein shake and follow storage, timing and preparation instructions
* Indicated by a qualified health care provider to safely participate in an exercise-based rehabilitation program
* Ability to read and comprehend the English language

Exclusion Criteria:

* Certain medical conditions, diagnosis, physical or psychological or physical exam finding that precludes participation, medications, or contraindications for protein supplement

  * Individuals who are determined by their health care provider to be contraindicated for participation in an exercise-based rehabilitation program
  * Individuals with food allergies to animal based products, nuts, and/or eggs
  * Individuals with consumption preferences omitting non-vegan or vegetarian products
  * Taking protein supplements already
  * History of severe liver disorder
  * History of Kidney disorder
  * History of diabetes
  * History of Gastrointestinal malabsorption
  * History of Parathyroid gland disorders
  * Pregnant, postpartum up to six months, lactating, or intention to become pregnant

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Muscle size | 3 months, 6 months, 1 year, 2 years
  Change in spine extensor muscle cross sectional area (cm2)

SECONDARY OUTCOMES:
Symptom inference - change in pain. Visual Analogue Scale (VAS), 0-100mm | 3 months, 6 months, 1 year, 2 years
  Difference in VAS (in mm) between initial evaluation and endpoint
Change in disability | 3 months, 6 months, 1 year, 2 years
  Difference in Oswestry Disability Index (ODI), between evaluation and end point
Patient Goal Achievement | 3 months, 6 months
  Patient Specific Functional Scale (PSFS), 0-10 points
Change in strength (lbs*deg) | 3 months, 6 months, 1 year, 2 years
  Difference in spine extension torque as measures by isokinetic dynamometer between initial evaluation and endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Shahidi, PT, PhD, Study Director — UCSD Orthopedic Surgery
Locations (1):
- SpineZone, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Patient data will only be accessible to SpineZone and collaborating research partners (UCSD).